CLINICAL TRIAL: NCT00426751
Title: Eptifibatide Versus Abciximab in Primary PCI for Acute ST Elevation Myocardial Infarction
Brief Title: Efficacy Of Eptifibatide Compared To Abciximab In Primary Percutaneous Coronary Intervention (PCI) For Acute ST Elevation Myocardial Infarction (STEMI)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 106915
Record Dates: First submitted 2007-01-24; First posted 2007-01-25 (Estimated); Results first posted 2010-04-26 (Estimated); Last update posted 2012-11-27 (Estimated); Status verified 2012-11

CONDITIONS: Infarction, Myocardial
Keywords: Eptifibatide; ST-elevation Myocardial Infarction; STEMI; Abciximab
MeSH Terms: conditions — Myocardial Infarction; ST Elevation Myocardial Infarction | interventions — Abciximab; Eptifibatide

ARMS (2):
- Abciximab (Active Comparator): Intravenous bolus of 0.25 mg/kg followed by continuous intravenous infusion of 0.125 mcg/kg/min (max. 10 mcg/min) for 12 h after PCI.
  Interventions: Drug: Abciximab
- Eptifibatide (Experimental): Intravenous bolus of 180 mcg/kg followed immediately by a continuous infusion of 2.0 mcg/kg/ min for 20-24 h after end of PCI, and a second bolus of 180 mcg/kg administered 10 min after the first bolus.
  Interventions: Drug: Eptifibatide

INTERVENTIONS:
Drug: Abciximab — Intravenous bolus of 0.25 mg/kg followed by continuous intravenous infusion of 0.125 mcg/kg/min (max. 10 mcg/min) for 12 h after PCI.
  Arms: Abciximab
Drug: Eptifibatide — Intravenous bolus of 180 mcg/kg followed immediately by a continuous infusion of 2.0 mdg/kg/ min for 20-24 h after end of PCI, and a second bolus of 180 mcg/kg administered 10 min after the first bolus.
  Other Names: Abciximab
  Arms: Eptifibatide

SUMMARY:
Multinational, multicentre, randomised, prospective, open, parallel group study directly comparing two glycoprotein-IIb/IIIa inhibitors, abciximab and eptifibatide, added early to standard treatment before primary PCI of STEMI patients with respect to effect on sum-ST-resolution after 60 minutes post-procedure and other measures of myocardial reperfusion

ELIGIBILITY:
Inclusion Criteria:

* Women must be postmenopausal (i.e.12 months without menstrual period), or surgically sterile, i.e. women of child bearing potential are not allowed to be included into the study. In cases of doubt a pregnancy test should be performed. (NB -post menopausal women currently receiving hormone replacement are permissible)
* Acute myocardial infarction < 12 h defined as:

  1. Angina or equivalent symptoms > 20 min and
  2. ST elevation in 2 contiguous ECG leads (= 2 mm precordial lead, = 1 mm limb lead). This ECG recording serves as baseline ECG, i.e. ECG I.
* Planned primary percutaneous coronary intervention
* The subject has given written informed, dated consent to participate in the study

Exclusion Criteria:

* Subjects not able to give informed consent
* Left Bundle Branch Block
* Thrombolytic therapy within 24 hours before randomization
* Oral anticoagulation with International Normalized Ratio (INR) > 2
* Known platelets < 100.000/µl or known hemorrhagic diathesis
* Stroke or Transient Ischemic Attack (TIA) within the past 6 months or any permanent residual neurological defect
* Evidence of an active gastrointestinal or urogenital bleeding
* Major surgery within 6 weeks
* History of allergic reaction to abciximab or eptifibatide or any component used in the study (including contrast media)
* Known severe renal (creatinine clearance <30ml/min) or hepatic insufficiency as well as Alanine transaminase (ALT)/aspartate transaminase (AST) elevations = 3xUpper limit normal (ULN); isolated AST-elevation is not considered an exclusion criteria from study participation
* Severe concomitant disease with life expectation < 1 year
* Subject has participated in any study using an investigational drug or device within 30 days or within 5 half-lives of the investigational drug (whichever is longer) of entry into this study.
* Subjects who will be inaccessible due to geographic or social factors during treatment or follow-up
* In France, a subject is neither affiliated with nor a beneficiary of a social security category.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 429 (Actual)
Dates: Start 2006-10; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (23):
- France (13):
  - GSK Investigational Site, Alençon
  - GSK Investigational Site, Bordeaux
  - GSK Investigational Site, Caen
  - GSK Investigational Site, Créteil
  - GSK Investigational Site, Lille
  - GSK Investigational Site, Melun
  - GSK Investigational Site, Nancy
  - GSK Investigational Site, Ollioules
  - GSK Investigational Site, Pau
  - GSK Investigational Site, Perpignan
  - GSK Investigational Site, Pessac
  - GSK Investigational Site, Toulon
  - GSK Investigational Site, Vandœuvre-lès-Nancy
- Germany (10):
  - GSK Investigational Site, Freiburg im Breisgau, Baden-Wurttemberg
  - GSK Investigational Site, Heidelberg, Baden-Wurttemberg
  - GSK Investigational Site, Würzburg, Bavaria
  - GSK Investigational Site, Offenbach, Hesse
  - GSK Investigational Site, Aachen, North Rhine-Westphalia
  - GSK Investigational Site, Dortmund, North Rhine-Westphalia
  - GSK Investigational Site, Mönchengladbach, North Rhine-Westphalia
  - GSK Investigational Site, Neuss, North Rhine-Westphalia
  - GSK Investigational Site, Ludwigshafen am Rhein, Rhineland-Palatinate
  - GSK Investigational Site, Homburg, Saarland

REFERENCES:
- [Derived] Zeymer U, Margenet A, Haude M, Bode C, Lablanche JM, Heuer H, Schroder R, Kropff S, Bourkaib R, Banik N, Zahn R, Teiger E. Randomized comparison of eptifibatide versus abciximab in primary percutaneous coronary intervention in patients with acute ST-segment elevation myocardial infarction: results of the EVA-AMI Trial. J Am Coll Cardiol. 2010 Aug 3;56(6):463-9. doi: 10.1016/j.jacc.2009.08.093. PMID 20670755

RESULTS

PARTICIPANT FLOW:
Groups:
- Eptifibatide: Intravenous bolus of 180 micrograms (µg)/kilogram (kg) Eptifibatide followed immediately by a continuous infusion of 2 µg/kg/minute (min) for 20-24 hours (hr) after the end of percutaneous coronary intervention (PCI), and a second bolus of 180 µg/kg administered 10 min after the first bolus
- Abciximab: Intravenous bolus of 0.25 mg/kg Abciximab followed by continuous intravenous infusion of 0.125 μg/kg/min (maximum 10 μg/min) for 12 hr after PCI
Period: Overall Study
Arm/Group | Eptifibatide | Abciximab
Started | 226 | 203
Completed | 204 | 183
Not Completed | 22 | 20
Not completed — Adverse Event | 8 | 1
Not completed — Lost to Follow-up | 7 | 6
Not completed — Consent Withdrawn | 0 | 1
Not completed — Other Reasons | 7 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Eptifibatide | Abciximab | Total
Number analyzed (Participants) | 214 | 196 | 410
Age Continuous [Mean (Standard Deviation); unit: years] — Twelve participants in the eptifibatide group and 6 participants in the abciximab group were excluded from the Intent-to-Treat (ITT) and Per Protocol (PP) Populations due to uncertain infarct localization. One of these participants in the abciximab group had not received study medication and was also excluded from safety analysis. One additional participant in the abciximab group had not received study medication and was also excluded from safety analysis.
  years | 61.3 (12.5) | 60.5 (12.7) | 60.9 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants] — Twelve participants in the eptifibatide group and 6 participants in the abciximab group were excluded from the Intent-to-Treat (ITT) and Per Protocol (PP) Populations due to uncertain infarct localization. One of these participants in the abciximab group had not received study medication and was also excluded from safety analysis. One additional participant in the abciximab group had not received study medication and was also excluded from safety analysis.
  Participants
    Female | 50 | 39 | 89
    Male | 164 | 157 | 321

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Complete Sum ST Resolution (STR) 60 Minutes (Min) After Percutaneous Coronary Intervention (PCI) (Per Protocol Population)
Description: Sum STR was calculated as the difference between baseline (ECG I) and ECG III. The sum STR is the segment elevation resolution from all ECG leads associated with the infarct location. ST resolution, a method used to evaluate myocardial reperfusion, was expressed as a percentage of the baseline value (Complete: ≥ 70% resolution).
Time Frame: Baseline (ECG I) and 60 min +/- 15 min after PCI (ECG III)
Population: Per Protocol (PP) Population: All randomized participants who received at least one dose of study drug, who had data that were fully evaluable for the primary endpoint, and who did not show any major protocol violation.
Measure: Number; unit: participants
Arm/Group | Eptifibatide | Abciximab
Number analyzed (Participants) | 113 | 111
participants | 71 | 65
Statistical Analysis 1: Comparison: Eptifibatide vs Abciximab; Test type: Non-Inferiority or Equivalence — For the assessment of differences between both treatment groups, a generalized model (under binomial probability distribution), adjusted for center, was applied; Median Difference (Final Values) = 2.1, 90% CI [-8.5 to 12.8]

2. Primary Outcome: Number of Participants With Complete Sum ST Resolution (STR) 60 Min After Percutaneous Coronary Intervention (PCI) (Intent-to-Treat Population)
Description: as for outcome 1
Time Frame: Baseline (ECG I) and 60 min +/- 15 min after PCI (ECG III)
Population: Intent-to-Treat (ITT) Population: All randomized participants who received at least one dose of study medication.
Measure: Number; unit: participants
Arm/Group | Eptifibatide | Abciximab
Number analyzed (Participants) | 214 | 196
participants | 124 | 103
Statistical Analysis 1: Comparison: Eptifibatide vs Abciximab; Test type: Non-Inferiority or Equivalence — For the assessment of differences between both treatment groups a generalised model (under binomial probability distribution), adjusted for centre, was applied; Mean Difference (Final Values) = 6.8, 95% CI [-3.0 to 16.6] — Analysis based on the ITT population confirmed the results observed in the PP population

3. Secondary Outcome: Number of Participants With Complete or Partial Sum ST Resolution (STR) 60 Min After PCI
Description: Sum STR was calculated as the difference between baseline (ECGI) and ECG III. The sum STR is the segment elevation resolution from all ECG leads associated with infarct location. ST resolution, a method used to evaluate myocardial reperfusion, was expressed as a percentage of the baseline (Complete: ≥ 70% resolution; Partial: ≥ 30% and < 70% resolution; None: < 30% resolution).
Time Frame: Baseline (ECG I) and 60 min +/- 15 min after PCI (ECG III)
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Eptifibatide | Abciximab
Number analyzed (Participants) | 214 | 196
participants
  Complete sum STR( ≥70%) | 124 | 103
  Complete or partial sum STR (≥30%) | 180 | 154
  Partial sum STR (≥30% and <70%) | 56 | 51
  No sum STR (<30%) | 34 | 42

4. Secondary Outcome: Number of Participants With Complete Single Lead ST Resolution (STR) 60 Min After PCI
Description: Single lead STR is calculated as the difference (as a percentage) between baseline (ECG I) and ECG III of either the ST elevation on one of the leads (II, III, aVF, V5, and V6) or the ST depression of one of the precordial leads (V1- V4), whichever lead showed the largest deviation either at baseline or at ECG III, respectively (Complete: ≥ 70%; Partial: ≥ 30% and <70%).
Time Frame: Baseline (ECG I) and 60 min +/- 15 min after PCI (ECG III)
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Eptifibatide | Abciximab
Number analyzed (Participants) | 214 | 196
participants | 105 | 82

5. Secondary Outcome: Mean Change From Baseline in the Sum ST Resolution 60 Min After PCI
Description: Sum STR was calculated as the difference between baseline (ECGI) and ECG III. The sum STR is the segment elevation resolution from all ECG leads associated with infarct location. ST resolution, a method used to evaluate myocardial reperfusion, was expressed as a percentage of the baseline.
Time Frame: Baseline (ECG I) and 60 min +/- 15 min after PCI (ECG III)
Population: ITT Population. Some participants were un-evaluable with regard to the primary endpoint and were counted as failures. These participants were excluded from this analysis.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Eptifibatide | Abciximab
Number analyzed (Participants) | 198 | 183
percent change | 71.6 (27.2) | 66.3 (31.1)

6. Secondary Outcome: Mean Change From Baseline in Single Lead ST Resolution (STR) 60 Min After PCI
Description: Single lead STR is calculated as the difference between baseline (ECG I) and ECG III of either the ST elevation on one of the leads (II, III, aVF, V5, and V6) or the ST depression of one of the precordial leads (V1 -V4), whichever lead showed the largest deviation either at baseline or at follow-up, respectively. STR was expressed as a percentage from baseline.
Time Frame: Baseline (ECG I) and 60 min +/- 15 min after PCI (ECG III)
Population: ITT Population. Participants with unevaluable ECGs were excluded from analysis.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Eptifibatide | Abciximab
Number analyzed (Participants) | 176 | 167
percent change | 70.2 (25.5) | 64.0 (28.7)

7. Secondary Outcome: Mean Change From Baseline in the Sum ST Resolution (STR) Before PCI
Description: Mean sum STR was calculated as the difference between baseline (ECGI) and ECG II: the mean of the sum of ST elevation resolution from all ECG leads associated with infarct location. ST resolution was expressed as a percentage from baseline.
Time Frame: Baseline (ECG I) and immediately prior to PCI (ECG II)
Population: ITT Population. Participants who did not have an ECG II immediately before PCI were excluded from analysis.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Eptifibatide | Abciximab
Number analyzed (Participants) | 145 | 120
percent change | 25.9 (32.0) | 21.2 (29.0)

8. Secondary Outcome: Mean Maximum ST Deviation Existing (Max STE) 60 Min After PCI
Description: Max STE is measured similarly to single-lead STR, but was not compared with the ST deviation on the baseline ECG I. It was the existing ST deviation on the single ECG lead of maximum ST deviation present at 60 minutes after the PCI (ECG III).
Time Frame: 60 min +/- 15 min after PCI (ECG III)
Population: ITT Population. Participants with unevaluable ECGs were excluded from analysis.
Measure: Mean (Standard Deviation); unit: millimeters (mm)
Arm/Group | Eptifibatide | Abciximab
Number analyzed (Participants) | 180 | 172
millimeters (mm) | 1.1 (1.1) | 1.4 (1.4)

9. Secondary Outcome: Number of Participants With the Indicated Patency of Infarcted Vessels According to Thrombolysis in Myocardial Infarction (TIMI) Classification Before PCI
Description: Number of participants with the respective patency of the infarcted vessels was evaluated by TIMI (Thrombolysis In Myocardial Infarction) flow grades (Grade 0 = No perfusion, Grade 1 = Penetration with minimal perfusion, Grade 2 = Partial perfusion, Grade 3 = Complete perfusion), as assessed by core angiography lab.
Time Frame: immediately before PCI
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Eptifibatide | Abciximab
Number analyzed (Participants) | 214 | 196
participants
  TIMI 3 patency before PCI | 74 | 59
  TIMI 2/3 patency before PCI | 85 | 67
  TIMI 0/1 patency before PCI | 117 | 123

10. Secondary Outcome: Number of Participants With TIMI 3 Patency of Infarcted Vessels Following PCI
Description: The number of participants with TIMI grade 3 (complete perfusion) patency of the infarcted vessels following PCI, as assessed by core angiography lab, was measured.
Time Frame: after PCI
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Eptifibatide | Abciximab
Number analyzed (Participants) | 214 | 196
participants | 145 | 137

11. Secondary Outcome: Mean Number of Corrected TIMI Frame Counts (cTIMI) Following PCI
Description: cTIMI frame counts (number of cineframes needed for dye to reach standardized distal landmarks in a coronary vessel; objective index of coronary blood flow) following PCI, as assessed by core angiography lab.
Time Frame: after PCI
Population: ITT Population. Participants with un-evaluable angiographies were excluded from analysis.
Measure: Mean (Standard Deviation); unit: number of frame counts
Arm/Group | Eptifibatide | Abciximab
Number analyzed (Participants) | 165 | 151
number of frame counts | 25.3 (21.0) | 23.6 (17.9)

12. Secondary Outcome: Number of Participants With the Indicated Myocardial Blush Grade (TIMI Myocardial Perfusion Grade [TMPG]) After PCI
Description: The number of participants with the indicated myocardial blush grade (TMPG), used to assess the myocardial reperfusion in the infarcted myocardium following PCI (as assessed by the core angiography laboratory), was measured. Blush grades: 0 = failure of dye to enter the microvasculature; 1 = dye slowly enters but fails to exit the microvasculature; 2 = delayed entry and exit of dye from the microvasculature; 3: normal entry and exit of dye from the microvasculature. Blush that is of only mild intensity throughout the washout phase but fades minimally is also classified as grade 3.
Time Frame: after PCI
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Eptifibatide | Abciximab
Number analyzed (Participants) | 214 | 196
participants
  Myocardial blush Grade 3 | 64 | 54
  Myocardial blush Grade 2 | 0 | 0
  Myocardial blush Grade 1 | 98 | 96
  Myocardial blush Grade 0 | 13 | 11
  Not assessable | 38 | 34

13. Secondary Outcome: Combined Endpoint: Number of Participants With Events of Death, Re-myocardial Infarction (MI), and Urgent Target Vessel Revascularisation (UTVR)
Description: The number of participants who died, experienced re-MI, or experienced UTVR (necessity of re-PCI of the target vessel or coronary artery bypass graft [CABG] because of recurrent ischaemic angina within 30 days after PCI) within the specified timeframe was measured.
Time Frame: Day 7 or hospital discharge; Day 30 after index-MI
Population: Safety Population: All participants who received at least one dose of study medication.
Measure: Number; unit: participants
Arm/Group | Eptifibatide | Abciximab
Number analyzed (Participants) | 226 | 201
participants
  Death, re-MI, or UTVR until day 7 or discharge | 12 | 14
  Death, re-MI, or UTVR until day 30 | 17 | 17

14. Secondary Outcome: Number of Participants Who Died, and/or Experienced Re-MI and UTVR (Individually Counted)
Description: The number of participants who died, and/or experienced re-MI or UTVR (individually counted) within the specified timeframe was measured.
Time Frame: Day 7 or hospital discharge; Day 30 after index-MI
Population: Safety Population
Measure: Number; unit: participants
Arm/Group | Eptifibatide | Abciximab
Number analyzed (Participants) | 226 | 201
participants
  Deaths until day 7 or discharge | 8 | 7
  Deaths until day 30 | 13 | 7
  Re-MI until day 7 or discharge | 0 | 3
  Re-MI until day 30 | 0 | 5
  UTVR until day 7 or discharge | 5 | 8
  UTVR until day 30 | 5 | 10

15. Secondary Outcome: Number of Participants Who Experienced Stroke or Major Bleeding Complications
Description: Number of participants who experienced stroke (hemorrhagic, non-hemorrhagic) or major bleedings (TIMI class: intracranial haemorrhage, spontaneous bleeding, bleeding at any instrumented site, retroperitoneal bleeding, or clinically significant overt haemorrhage associated with a drop in haematocrit of ≥ 15% or a drop in haemoglobin of ≥ 5 g/dL).
Time Frame: Day 7 or hospital discharge; Day 30 after index-MI
Population: Safety Population
Measure: Number; unit: participants
Arm/Group | Eptifibatide | Abciximab
Number analyzed (Participants) | 226 | 201
participants
  Stroke or major bleeding until day 7 or discharge | 6 | 1
  Stroke or major bleeding until day 30 | 6 | 2

16. Secondary Outcome: Number of Participants Who Died and or Experienced Re-MI Until 6 Months After PCI
Description: The number of participants who died and/or experienced re-MI within 6 month after PCI was measured.
Time Frame: until 6 Month (Day 180) after index-MI
Population: Safety Population
Measure: Number; unit: participants
Arm/Group | Eptifibatide | Abciximab
Number analyzed (Participants) | 226 | 201
participants | 15 | 15

17. Secondary Outcome: Number of Participants With Heart Failure Until 6 Months After PCI
Description: The number of participants with heart failure within 6 month after PCI was measured.
Time Frame: until 6 Months (Day 180) after index-MI
Population: Safety Population
Measure: Number; unit: participants
Arm/Group | Eptifibatide | Abciximab
Number analyzed (Participants) | 226 | 201
participants | 23 | 22

18. Secondary Outcome: Number of Participants With Major Bleedings (TIMI Classification)
Description: Number of participants with major bleedings (according to TIMI classification: intracranial haemorrhage, spontaneous bleeding, bleeding at any instrumented site, retroperitoneal bleeding, or clinically significant overt haemorrhage associated with a drop in haematocrit of ≥ 15% or a drop in haemoglobin of ≥ 5 g/dL) within the specified timeframe was measured.
Time Frame: Day 7 or hospital discharge; Day 30 after index-MI
Population: Safety Population
Measure: Number; unit: participants
Arm/Group | Eptifibatide | Abciximab
Number analyzed (Participants) | 226 | 201
participants
  Major bleedings (TIMI classification) until day 7 | 6 | 0
  Major bleedings (TIMI classification) until day 30 | 6 | 1

19. Secondary Outcome: Number of Participants With Minor Bleedings (TIMI Classification)
Description: The number of participants with minor bleedings (according to TIMI classification: clinically overt bleeding [e.g., gross haematuria or haematemesis) associated with a drop in haematocrit of ≥ 9% or a drop in haemoglobin of ≥ 3 g/dL) within the specified timeframe was measured.
Time Frame: Day 7 or hospital discharge; Day 30 after index-MI
Population: Safety Population
Measure: Number; unit: participants
Arm/Group | Eptifibatide | Abciximab
Number analyzed (Participants) | 226 | 201
participants
  Minor bleedings (TIMI classification) until day 7 | 19 | 12
  Minor bleedings (TIMI classification) until day 30 | 19 | 12

20. Secondary Outcome: Mean Duration of Stay in the Ward
Description: Costs were measured as the duration of stay in the ward (outpatient, normal ward, and intensive care unit) within the specified timeframe was measured.
Time Frame: until 6 months after index-MI
Population: ITT Population
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Eptifibatide | Abciximab
Number analyzed (Participants) | 211 | 195
days | 8.0 (6.7) | 9.7 (11.9)

ADVERSE EVENTS:
Arm/Group | Eptifibatide | Abciximab
Serious Adverse Events (participants affected / at risk) | 24/226 | 19/201
Other Adverse Events (participants affected / at risk) | 49/226 | 28/201
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eptifibatide (N=226) | Abciximab (N=201)
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 2 | 2
Atrioventricular block complete (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 2 | 0
Cardiogenic shock (Cardiac disorders) | 4 | 2
In-stent coronary artery restenosis (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 2
Ventricular fibrillation (Cardiac disorders) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 2 | 0
Ventricular septal defect (Congenital, familial and genetic disorders) | 0 | 1
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 0
General physical health deterioration (General disorders) | 1 | 0
Malaise (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 1
Sudden death (General disorders) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Gastrointestinal infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 1
Sepsis (Infections and infestations) | 0 | 1
Staphylococcal infection (Infections and infestations) | 0 | 1
Tracheobronchitis (Infections and infestations) | 0 | 1
Coronary artery reocclusion (Injury, poisoning and procedural complications) | 1 | 0
In-stent arterial restenosis (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Intervertebral disc displacement (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebral hemorrhage (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Testicular pain (Reproductive system and breast disorders) | 1 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Aortic dissection (Vascular disorders) | 1 | 0
Haemorrhage (Vascular disorders) | 2 | 0
Shock (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Eptifibatide (N=226) | Abciximab (N=201)
Angina pectoris (Cardiac disorders) | 11 | 5
Cardiac failure (Cardiac disorders) | 5 | 0
Ventricular extrasystoles (Cardiac disorders) | 7 | 4
Ventricular tachycardia (Cardiac disorders) | 9 | 6
Post procedural heamatoma (Injury, poisoning and procedural complications) | 12 | 9
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 0
Headache (Nervous system disorders) | 0 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.